CLINICAL TRIAL: NCT02206945
Title: Neurofeedback of Activity in the Orbitofrontal Cortex for OCD
Brief Title: Neurofeedback for Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0206017435-2; R01MH100068 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- neurofeedback (Experimental): Two imaging sessions of neurofeedback.
  Interventions: Behavioral: neurofeedback
- control feedback (Placebo Comparator): Two imaging sessions of feedback
  Interventions: Behavioral: control feedback

INTERVENTIONS:
Behavioral: neurofeedback — Subject provided with feedback of activity in target brain area in the form of a line graph. Cued to try to make the line go up at certain times and down at other times.
  Arms: neurofeedback
Behavioral: control feedback — Subject provided with a control/placebo type of feedback in the form of a line graph. Cued to try to make the line go up at certain times and down at other times.
  Arms: control feedback

SUMMARY:
The aim of this study is to train patients with obsessive-compulsive disorder to control a region of their brain that has been associated with their symptoms. Patients in the experimental group will be given direct feedback regarding activity in this brain area while they are undergoing functional magnetic resonance imaging (fMRI) scanning, and will try to learn to control activity in the region during these feedback sessions. A separate group of patients will be given a control form of feedback that we do not believe can have clinical benefits. Our primary hypothesis is that the neurofeedback training will reduce OCD symptoms more than the control feedback.

DETAILED DESCRIPTION:
Original study design recruiting controls who were matched to the experimental group was changed to a randomized design prior to enrollment of the first participant.

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnosis of Current OCD, based on Diagnostic and Statistical Manual (DSM-IV) criteria, a Y-BOCS (Yale-Brown Obsessive-Compulsive Scale) score >=16
* Principle OCD symptoms- Primary symptoms must be either Cleaning/Contamination or Checking; other symptoms okay
* Unmedicated (or medications stable for 8 weeks).
* Research group must be able to identify a target region in the orbitofrontal cortex that is related to symptoms

Exclusion Criteria:

* Active Psychosis; Pervasive Developmental Disorder ; epilepsy or other major neurological disorder
* History of major head trauma or psychosurgery
* Active Substance Abuse within 6 months
* Seizure disorder or other significant neurological disorder
* Active Suicidality
* Pregnancy
* severe claustrophobia, ferromagnetic metal in the body, a pacemaker or defibrillator, or any other condition that would make MRI scanning unsafe or inappropriate
* any psychotropic medication other than a selective serotonin reuptake inhibitor (SSRI) antidepressant, anafranil, or a low-dose hypnotic or anxiolytic taken on an as-needed basis
* active cognitive/behavioral therapy initiated within the last 3 months (continuation of established maintenance therapy that has been going on for longer than 3 months will not be grounds for exclusion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07; Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
A modified version of the Yale-Brown Obsessive-Compulsive Symptom scale (Y-BOCS) will be used, that queries subjects regarding symptoms | Immediately before intervention
A modified version of the Yale-Brown Obsessive-Compulsive Symptom scale (Y-BOCS) will be used, that queries subjects regarding symptoms | Approximately 4 days post-intervention

SECONDARY OUTCOMES:
Control over target brain area | Approximately 4 days pre-intervention
  Control task scans will be conducted in which subjects are cued to at times to increase activity in their target brain area and at other times to decrease activity in their target brain area. During both conditions they will be presented with symptom provoking images. The percent signal change in the BOLD signal in the target area during increase relative to decrease blocks will be used as the measure of control over the brain area.
Control over the target brain area. | Approximately 4 days post-intervention
  Control task scans will be conducted in which subjects are cued to at times to increase activity in their target brain area and at other times to decrease activity in their target brain area. During both conditions they will be presented with symptom provoking images. The percent signal change in the BOLD signal in the target area during increase relative to decrease blocks will be used as the measure of control over the brain area.

OTHER OUTCOMES:
Functional connectivity patterns in the brain | Approximately 4 days pre-intervention
  Functional connectivity will be assessed based on temporal correlations in resting state functional imaging data.
Functional connectivity patterns in the brain | Approximately 4 days post-intervention
  Functional connectivity will be assessed based on temporal correlations in resting state functional imaging data.
A modified version of the Yale-Brown Obsessive-Compulsive Symptom scale (Y-BOCS) will be used, that queries subjects regarding symptoms | Approximately 2 weeks post-intervention
A modified version of the Yale-Brown Obsessive-Compulsive Symptom scale (Y-BOCS) will be used, that queries subjects regarding symptoms | Approximately 4 weeks post-intervention
Average self-report of washing/checking anxiety to provocative images during a session in which they are instructed to control anxiety | Approximately 4 days pre-intervention
  Subject instructed to control anxiety, shown provocative pictures and self-reports the anxiety they experience for each image. Responses averaged over session for a single number representing level of anxiety experienced despite efforts to control that anxiety.
Average self-report of washing/checking anxiety to provocative images during a session in which they are instructed to control anxiety. | Approximately 4 days post-intervention
  Subject instructed to control anxiety, shown provocative pictures and self-reports the anxiety they experience for each image. Responses averaged over session for a single number representing level of anxiety experienced despite efforts to control that anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hampson, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Rance M, Zhao Z, Zaboski B, Kichuk SA, Romaker E, Koller WN, Walsh C, Harris-Starling C, Wasylink S, Adams T Jr, Gruner P, Pittenger C, Hampson M. Neurofeedback for obsessive compulsive disorder: A randomized, double-blind trial. Psychiatry Res. 2023 Oct;328:115458. doi: 10.1016/j.psychres.2023.115458. Epub 2023 Sep 3. PMID 37722238